CLINICAL TRIAL: NCT02938806
Title: The Effects of Type 1 Diabetes Mellitus and Increased Weight on Gut Microbiome and Urine Metabolome Profiles in Children
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr Jane Kim, Assistant Professor, University of California, San Diego
Other Study IDs: #160113
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Overweight; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Obese/overweight children with T1D: No intervention
  Interventions: Other: No intervention
- Normal weight children with T1D: No intervention
  Interventions: Other: No intervention
- Obese/overweight children, no diabetes: No intervention
  Interventions: Other: No intervention
- Healthy, normal weight children: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study employs a cross-sectional design to profile the gut microbiome and urine metabolome in overweight/obese children with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
The investigators will obtain stool and urine samples from subjects aged 7-17 years in 4 groups:

* Group 1: Obese or overweight children within 3 years of diagnosis of T1D
* Group 2: Normal weight children within 3 years of diagnosis of T1D
* Group 3: Obese or overweight children without T1D
* Group 4: Normal weight children without T1D

Type 1 diabetes will be defined according to American Diabetes Association criteria along with the presence of pancreatic autoantibodies (GAD65, ICA512, or insulin autoantibodies). Obese and overweight status will be defined by BMI >85th percentile for age and gender according to CDC criteria.

All subjects will provide one-time stool and first morning urine sample. Overweight or obese subjects will additionally have a point of care blood glucose and hemoglobin A1c measurement to ensure that they do not have diabetes.

The investigators will perform 16S rRNA sequencing of stool bacteria and mass spectrometry measurement of urine metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 to 17 years
* Diagnosis of diabetes will be defined by current American Diabetes Association criteria ° (fasting glucose > 126 mg/dl, 2 hour OGTT glucose > 200 mg/dl; random glucose > 200 with symptoms of hyperglycemia; or HbA1c > 6.5%)
* Diabetes duration < 3 years
* Presence of pancreatic autoimmunity (GAD65, ICA512, or insulin autoantibody positivity)
* Adult caregiver willing to actively support study participation
* Signed parental informed consent form and minor child informed assent form

Exclusion Criteria:

* Other significant organ system illness or condition (including psychiatric or developmental disorder) that, in the opinion of the investigator, would prevent participation

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 7-17 years with/without T1DM and with/without obese/overweight status in San Diego, California
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-06; Primary Completion 2019-04 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Analysis of gut microbial composition and diversity by 16S rRNA sequencing | 2 years

SECONDARY OUTCOMES:
Analysis of urine metabolite concentrations measured by mass spectrometry | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kim, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Rady Children's Hospital Endocrinology Department, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boerner BP, Sarvetnick NE. Type 1 diabetes: role of intestinal microbiome in humans and mice. Ann N Y Acad Sci. 2011 Dec;1243:103-18. doi: 10.1111/j.1749-6632.2011.06340.x. PMID 22211896
- [Background] Dunne JL, Triplett EW, Gevers D, Xavier R, Insel R, Danska J, Atkinson MA. The intestinal microbiome in type 1 diabetes. Clin Exp Immunol. 2014 Jul;177(1):30-7. doi: 10.1111/cei.12321. PMID 24628412
- [Background] Zimny D, Szatkowska M, Polubok J, Maciaszek J, Machaj M, Barg E. [The use of metabolomics in medicine - some examples of oncological and metabolic diseases]. Pediatr Endocrinol Diabetes Metab. 2015;20(2):55-62. doi: 10.18544/PEDM-20.02.0003. Polish. PMID 26615014